CLINICAL TRIAL: NCT03529617
Title: Pharmacokinetics of Liposomal Amphotericin B in Critically Ill vs. Non-critically Ill Hematological Patients: Exploration of Covariates
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S59273
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pharmacokinetics; Liposomal Amphotericin B; Critically Ill Patients
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Blood (plasma) Urine BAL (bronchoalveolar lavage) Ascitic fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Critically ill patients: Patients admitted on ICU.
  Interventions: Other: Sample collection
- Hematology patients: Patients admitted on the hematology ward.
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Plasma, urine, BAL and ascitic fluid sample collection.

SUMMARY:
This prospective study will compare the pharmacokinetic exposure to liposomal amphotericin B between critically ill patients and non-critically ill (hematology) patients in an early and late exposure day.

DETAILED DESCRIPTION:
This phase IV, open label, non-randomized, monocenter pharmacokinetic study will be carried out in critically ill and non-critically ill (hematology) patients receiving multiple dose treatment with L-AmB.

The pharmacokinetic exposure to liposomal amphotericin B in plasma, urine, BAL and ascitic fluid will be compared between the two population groups in an early and late exposure day.

Correlating covariates will be identified to provide a rationale for optimal dosing strategy in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with L-AmB
* Admitted to an ICU or Hematology ward

Exclusion Criteria:

* DNR 2 or 3
* Pregnant or lactating women
* Previous documentation of intolerance/sensitivity to L-AmB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. critically ill patients treated with L-AmB
  2. hematology patients treated with L-AmB
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma exposure and PK parameters | July 2020
  To document and compare plasma exposure and PK parameters in an ICU vs. non ICU hematology patient cohort in the early and late phase of L-AmB treatment.

SECONDARY OUTCOMES:
Covariates | July 2020
  To document correlating covariates and to stimulate the pharmacokinetics of L-AmB to provide a rationale for optimal dosing strategy in critically ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided